CLINICAL TRIAL: NCT02317887
Title: A Phase I/IIa Study of RS1 Ocular Gene Transfer for X-linked Retinoschisis
Brief Title: Study of RS1 Ocular Gene Transfer for X-linked Retinoschisis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VegaVect, Inc. (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15EI0038; 15-EI-0038 (Other Grant/Funding Number: National Eye Institute (NEI))
Record Dates: First submitted 2014-12-16; First posted 2014-12-17 (Estimated); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Retinoschisis; X-Linked
Keywords: Gene Transfer; X-Linked; Retinoschisis; AAV Vector
MeSH Terms: conditions — Retinoschisis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): 1e9 vg/eye
  Interventions: Biological: RS1 AAV Vector
- Cohort 2 (Experimental): 1e10 vg/eye
  Interventions: Biological: RS1 AAV Vector
- Cohort 3 (Experimental): 1e11 vg/eye
  Interventions: Biological: RS1 AAV Vector
- Cohort 4 (Experimental): 1e11 vg/eye
  Interventions: Biological: RS1 AAV Vector
- Cohort 5 (Experimental): 3e11 vg/eye
  Interventions: Biological: RS1 AAV Vector
- Cohort 6 (Experimental): Not to exceed 6e11 vg/eye
  Interventions: Biological: RS1 AAV Vector

INTERVENTIONS:
Biological: RS1 AAV Vector — Gene transfer by intravitreal injection of the RS1 AAV vector (AAV8-scRS/IRBPhRS)

SUMMARY:
Background:

- X-linked juvenile retinoschisis (XLRS) is caused by changes in the RS1 gene. These changes cause abnormal function of the eye protein retinoschisin. Without normal retinoschisin, the layers of the retina split and vision is lost. Researchers want to try to introduce a healthy RS1 gene into eye cells, to see if this helps retinal cells make healthy retinoschisin. They will put the gene in a virus. The gene and virus package is known as a gene transfer vector (AAV-RS1 vector).

Objectives:

- To see if the AAV-RS1 vector is safe to use in patients with X-linked retinoschisis.

Eligibility:

- Adults 18 and older with a mutation of the RS1 gene, 20/63 vision or worse in one eye, and XLRS.

Design:

* Participants will be screened with genetic tests to confirm XLRS. They will have a medical history and physical and eye exams.
* At visits 1-2, participants will have some or all of the following:
* Medical history
* Physical exam
* Blood and urine tests
* Tuberculosis skin test
* Eye exam
* Vision tests (for one test an intravenous line will be placed in the arm. A dye will be injected that will travel to the blood vessels in the eye).
* At visit 3, the AAV-RS1 vector will be injected with a needle in the study eye. Participants pupils will be dilated. They will get numbing eye drops.
* Visits 4-13 will occur in the 18 months after gene transfer. Many of the above tests will be repeated. Participants will discuss any side effects.
* Visits 14-17 will occur yearly between years 2 and 5.
* After year 5, participants will be contacted yearly by phone for up to 15 years.

DETAILED DESCRIPTION:
Objective: To evaluate the safety and tolerability of ocular AAV-RS1 vector (AAV8-scRS/IRBPhRS) gene transfer to the retina of participants affected with X-linked juvenile retinoschisis (XLRS).

Study Population: Male participants affected with XLRS will receive ocular gene transfer. A maximum of up to 24 participants may be enrolled.

Design: This is a Phase I/IIa, prospective, dose escalation, single-center study. One eye of each participant will receive the AAV-RS1 gene vector application by intravitreal injection. Participants will be closely monitored in conjunction with DSMC oversight. Participants will be followed for 18 months after which they will continue to be followed for up to 5 years after enrollment, or per FDA requirements, for further safety analysis.

Outcome Measures: The primary outcome is the safety of ocular AAV-RS1 vector as determined from assessment of retinal function, ocular structure and occurrence of adverse events and laboratory tests. Secondary outcomes include changes in visual function, electroretinogram (ERG) responses, visual field measurements, retinal imaging with optical coherence tomography (OCT), and the formation of anti-AAV and anti-RS1 antibodies.

Statistics: No formal sample size calculations are used in this Phase I/IIa dose-escalation study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participant is male with a mutation in the RS1 gene identified by genotyping.
* Participant must be 18 years of age or older.
* Participant must be able to understand and sign the informed consent.
* Participant must be medically able to comply with the study treatment, study testing and procedures and follow-up visits.
* Participant has at least one eye that meets the study eye criteria listed below.
* Participant must agree to use effective barrier (male or female condom) of contraception starting two weeks before and continuing one year after gene transfer.
* If the participant's partner is able to become pregnant, a second form of effective contraception will be required starting two weeks before and continuing one year after gene transfer.

Effective methods of contraception for this study include:

* hormonal contraception (birth control pills, injected hormones or vaginal ring),
* intrauterine device,
* barrier methods (condom or diaphragm) combined with spermicide,
* surgical sterilization (hysterectomy or tubal ligation in partner or vasectomy).

EXCLUSION CRITERIA:

* Participant is actively receiving another study medication/investigational product (IP).
* Participant has previously enrolled in another gene therapy trial.
* Participant is currently taking, or has taken in the last three months, a systemic carbonic anhydrase inhibitor prior to enrollment/baseline 1 testing.
* Participant has any condition that significantly increases risk of systemic corticosteroids or systemic steroid-sparing immuno-modulatory agents, such as HIV, syphilis, tuberculosis, hepatitis B, hepatitis C, or diabetes mellitus (DM).
* Participant has an underlying serious illness that impairs regular follow-up during the study.
* Participant has had diagnosis or treatment of a malignancy (excluding non-melanoma skin cancer) within the previous five years.
* Participant has pre-existing ocular tumors (excluding non-suspicious nevi).
* Participant has a known allergy to fluorescein dye or other contraindications to obtaining a fluorescein angiogram.
* Participant is on a medication that prevents safe administration of study related drugs.
* Participant has uncontrolled hypertension. (Hypertension judged to be adequately controlled at baseline medical evaluation is not exclusionary.)
* Participant has compromised renal function such that cyclosporine or Cellcept, which could be used to treat any manifest ocular inflammation, would be contraindicated.
* Participant has significant liver disease with elevated liver enzymes (greater than or equal to 2.5 times upper limit of normal [ULN]).
* Participant has low absolute neutrophil count (ANC<1.3 x 10(3)/micro liters).
* Participant has used any biologic immunosuppressive agents within the last three months (within the last six months for rituximab or cyclophosphamide).

STUDY EYE ELIGIBILITY CRITERIA:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

STUDY EYE INCLUSION CRITERIA:

* The study eye must have a best-corrected E-ETDRS visual acuity letterscore of less than or equal to 63 (i.e., worse than or equal to 20/63). The visual acuity from the first baseline visit (Baseline 1) will be used for eligibility determination in case of a change in visual acuity at the second baseline visit (Baseline 2).
* Electroretinogram in the study eye with a scotopic combined response demonstrating a subnormal b wave, consistent with retinoschisis.

STUDY EYE EXCLUSION CRITERIA:

* The study eye has a history of other ocular disease likely to contribute significantly to visual loss or likely to present special risks (e.g., optic neuropathy, advanced glaucoma, uveitis, large bullous schisis cavities or bullous retinal detachment precluding safe intravitreal injection).
* The study eye has lens, cornea, or other media opacities precluding adequate visualization and testing of the retina.
* The study eye has undergone intraocular surgery within six months prior to enrollment.
* The study eye is receiving topical carbonic anhydrase inhibitor, or has received topical carbonic anhydrase inhibitors in the past three months.

STUDY EYE SELECTION CRITERIA:

If both eyes of a participant meet the study eye eligibility criteria, the choice of study eye will be determined as follows:

* The eye with the worse visual acuity will be selected as the study eye.
* If both eyes have visual acuities within five letter differences of one another, the choice of study eye will be determined at the discretion of the Investigator in consultation with the participant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laryssa A Huryn, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vijayasarathy C, Zeng Y, Marangoni D, Dong L, Pan ZH, Simpson EM, Fariss RN, Sieving PA. Targeted Expression of Retinoschisin by Retinal Bipolar Cells in XLRS Promotes Resolution of Retinoschisis Cysts Sans RS1 From Photoreceptors. Invest Ophthalmol Vis Sci. 2022 Oct 3;63(11):8. doi: 10.1167/iovs.63.11.8. PMID 36227606
- [Derived] Vijayasarathy C, Sardar Pasha SPB, Sieving PA. Of men and mice: Human X-linked retinoschisis and fidelity in mouse modeling. Prog Retin Eye Res. 2022 Mar;87:100999. doi: 10.1016/j.preteyeres.2021.100999. Epub 2021 Aug 11. PMID 34390869
- [Derived] Mishra A, Vijayasarathy C, Cukras CA, Wiley HE, Sen HN, Zeng Y, Wei LL, Sieving PA. Immune function in X-linked retinoschisis subjects in an AAV8-RS1 phase I/IIa gene therapy trial. Mol Ther. 2021 Jun 2;29(6):2030-2040. doi: 10.1016/j.ymthe.2021.02.013. Epub 2021 Feb 15. PMID 33601057
- [Derived] Cukras C, Wiley HE, Jeffrey BG, Sen HN, Turriff A, Zeng Y, Vijayasarathy C, Marangoni D, Ziccardi L, Kjellstrom S, Park TK, Hiriyanna S, Wright JF, Colosi P, Wu Z, Bush RA, Wei LL, Sieving PA. Retinal AAV8-RS1 Gene Therapy for X-Linked Retinoschisis: Initial Findings from a Phase I/IIa Trial by Intravitreal Delivery. Mol Ther. 2018 Sep 5;26(9):2282-2294. doi: 10.1016/j.ymthe.2018.05.025. Epub 2018 Jul 7. PMID 30196853
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-EI-0038.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Started | 3 | 3 | 3 | 2 | 1 | 0
Completed | 3 | 3 | 3 | 2 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled into Cohort 6.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 1 | 0 | 12
Number analyzed (Eyes) | 6 | 6 | 6 | 4 | 2 | 0 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 3 | 2 | 1 | 0 | 11
  >=65 years | 1 | 0 | 0 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (11.5) | 47.7 (11.9) | 36.3 (12.2) | 41.0 (5.7) | 38.0 |  | 45.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 |  | 0
  Male | 3 | 3 | 3 | 2 | 1 |  | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 |  | 2
  Not Hispanic or Latino | 2 | 3 | 3 | 2 | 0 |  | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 0 | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 |  | 0
  White | 3 | 3 | 3 | 2 | 1 |  | 12
  More than one race | 0 | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 2 | 1 |  | 12
Electroretinography Combined Response Amplitudes [Mean (Standard Deviation); unit: µv] — The higher the amplitude, the better. Taken as the average of baseline 1 and 2 measurements. Population: Each individual measure summarizes data at the eye-level (either Study Eye or Fellow Eye) as indicated in the description of the measure itself.
  µv
    number analyzed (Eyes) | 3 | 3 | 3 | 2 | 1 | 0 | 12
    Dark-Adapted Rod Amplitude: Study Eye | 51.5 (40.7) | 64.7 (34.6) | 57.2 (8.7) | 75.0 (25.5) | 130.0 |  | 66.7 (32.5)
    Dark-Adapted Rod Amplitude: Fellow Eye | 73.8 (50.2) | 46.3 (4.8) | 70.3 (31.5) | 73.8 (14.5) | 149.5 |  | 72.4 (37.3)
    Dark-Adapted Combined Rod-Cone A-Wave 0dB Amplitude: Study Eye | 166.8 (38.6) | 222.5 (48.0) | 201.3 (17.5) | 162.5 (8.5) | 211.5 |  | 192.4 (37.3)
    Dark-Adapted Combined Rod-Cone A-Wave 0dB Amplitude: Fellow Eye | 180.2 (60.8) | 176.5 (75.8) | 190.5 (21.9) | 186.8 (23.7) | 235 |  | 187.5 (45.9)
    Dark-Adapted Combined Rod-Cone B-Wave 0dB Amplitude: Study Eye | 122.5 (60.7) | 175.2 (22.8) | 142.5 (17.1) | 125.8 (34.3) | 243.0 |  | 151.3 (47.0)
    Dark-Adapted Combined Rod-Cone B-Wave 0dB Amplitude: Fellow Eye | 138.2 (66.6) | 134.3 (21.6) | 138.2 (24.8) | 137.25 (42.1) | 294 |  | 150.0 (56.8)
    Dark-Adapted Combined Rod-Cone A-Wave 11dB Amplitude: Study Eye | 260.0 (46.8) | 298.5 (57.0) | 297.0 (17.5) | 258.3 (34.3) | 272.5 |  | 279.6 (39.0)
    Dark-Adapted Combined Rod-Cone A-Wave 11dB Amplitude: Fellow Eye | 276.2 (89.0) | 244.8 (96.2) | 259.5 (15.1) | 269.8 (64.0) | 301.5 |  | 265.2 (61.8)
    Dark-Adapted Combined Rod-Cone B-Wave 11dB Amplitude: Study Eye | 175.0 (67.2) | 202.5 (19.3) | 193.3 (10.9) | 175.0 (62.2) | 288.0 |  | 195.9 (47.4)
    Dark-Adapted Combined Rod-Cone B-Wave 11dB Amplitude: Fellow Eye | 197.8 (73.3) | 171.5 (15.5) | 184.3 (23.3) | 184.8 (64.0) | 313.0 |  | 195.3 (54.4)
    Dark-Adapted Oscillatory Potentials Amplitude: Study Eye | 13.8 (7.3) | 25.2 (11.0) | 19.3 (12.4) | 23.3 (15.2) | 46.0 |  | 22.3 (12.5)
    Dark-Adapted Oscillatory Potentials Amplitude: Fellow Eye | 13.7 (5.4) | 19.5 (5.6) | 22.2 (18.6) | 26.5 (20.5) | 61.5 |  | 23.4 (16.6)
    Light-Adapted Cone B-Wave 0dB Amplitude: Study Eye | 39.3 (23.6) | 66.2 (22.8) | 60.7 (14.5) | 62.5 (41.0) | 97.5 |  | 60.1 (25.4)
    Light-Adapted Cone B-Wave 0dB Amplitude: Fellow Eye | 46.8 (22.5) | 57.8 (13.7) | 66.3 (23.3) | 75.0 (48.8) | 106.0 |  | 64.1 (26.8)
    Light-Adapted Cone A-Wave 11dB Amplitude: Study Eye | 57.2 (10.1) | 75.5 (13.7) | 76.5 (8.5) | 68.5 (14.1) | 66.5 |  | 69.3 (12.2)
    Light-Adapted Cone A-Wave 11dB Amplitude: Fellow Eye | 59.2 (23.3) | 66.5 (9.6) | 70.7 (23.9) | 65.5 (24.7) | 63.0 |  | 65.3 (17.2)
    Light-Adapted Flicker Amplitude: Study Eye | 33.8 (15.3) | 55.8 (25.3) | 46.2 (11.5) | 55.8 (25.8) | 76.0 |  | 49.6 (19.9)
    Light-Adapted Flicker Amplitude: Fellow Eye | 37.5 (12.1) | 47.8 (13.3) | 52.7 (26.6) | 63.0 (38.2) | 82.5 |  | 51.9 (22.1)
Best Corrected Visual Acuity [Mean (Standard Deviation); unit: letters read] — Best corrected visual acuity (BCVA) as measured via Electronic Visual Acuity (EVA). Taken as the average of baseline 1 and 2 measurements. Population: Each individual measure summarizes data at the eye-level (either Study Eye or Fellow Eye) as indicated in the description of the measure itself.
  letters read
    number analyzed (Eyes) | 3 | 3 | 3 | 2 | 1 | 0 | 12
    Study Eye | 43.7 (8.5) | 45.8 (16.5) | 48.7 (8.4) | 52.0 (2.8) | 61.0 |  | 48.3 (10.0)
    Fellow Eye | 51.8 (4.9) | 59.5 (6.9) | 66.2 (4.1) | 66.3 (8.8) | 68.0 |  | 61.1 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs) Affecting Ocular Function That Differ Clinically From Those Expected in the Normal Course of Progression of XLRS
Description: Includes a) substantial functional change (change >=10 electronic visual acuity letters in best-corrected visual acuity from average of baseline visits), b) decrease in electroretinogram response amplitude (>=75% from average of baseline visits), c) severe ocular inflammation beyond inflammation anticipated consequent to an intravitreal injection; d) adverse events deemed clinically-related to the intraocular administration technique, and e) abnormal laboratory findings beyond Grade 1 Common Terminology Criteria for Adverse Events v5.0 and/or clinically significantly different than baseline. a)-d) only includes events occurring in the study eye.
Time Frame: Day 0 through Year 2, inclusive
Population: Includes all participants enrolled in the study and were administered the AAV vector injection, regardless of follow-up.
Measure: Number; unit: events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 1 | 0
events
  AEs affecting ocular function (differ clinically from expected in normal progression of XLRS) | 3 | 3 | 12 | 6 | 30 |
  Substantial functional change (Day 0-Year 2) | 0 | 0 | 3 | 0 | 21 |
  Decrease in Electroretinogram Response Amplitude (Day 0-Year 2) | 0 | 0 | 0 | 0 | 0 |
  Severe Ocular Inflammation (Day 8-Year 2) | 0 | 0 | 0 | 0 | 0 |
  AEs Clinically Related to Intraocular Administration Technique (Day 8-Year 2) | 0 | 2 | 8 | 2 | 9 |
  Abnormal Laboratory Findings (Day 0-Year 2) | 3 | 1 | 1 | 4 | 0 |

2. Secondary Outcome: Change in Electroretinography Combined Response Amplitudes
Description: Change in electroretinography combined response amplitudes from average of baseline 1 and 2 measurements. The higher the amplitude, the better.
Time Frame: Baseline 1 through Year 2
Population: Includes all participants enrolled in the study and were administered the AAV vector injection, regardless of follow-up with data available for at least one baseline visit and at Year 2.
Measure: Mean (Standard Deviation); unit: µV
Units Other Than Participants: Eyes
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 1 | 0
Number analyzed (Eyes) | 6 | 6 | 6 | 2 | 2 | 0
µV
  Dark-Adapted Rod Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Rod Amplitude: Study Eye | 13.8 (19.3) | -21.7 (13.5) | -13.8 (16.2) | -19.0 | -11.0 |
  Dark-Adapted Rod Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Rod Amplitude: Fellow Eye | -8.5 (25.5) | 14.0 (45.2) | -14.0 (38.5) | 4.5 | 14.5 |
  Dark-Adapted Combined Rod-Cone A-Wave 0dB Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Combined Rod-Cone A-Wave 0dB Amplitude: Study Eye | -0.5 (40.3) | -45.5 (19.5) | -21.7 (23.0) | 15.5 | -15.5 |
  Dark-Adapted Combined Rod-Cone A-Wave 0dB Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Combined Rod-Cone A-Wave 0dB Amplitude: Fellow Eye | -20.8 (10.4) | -21.8 (19.5) | -7.5 (6.8) | 4.5 | -2.0 |
  Dark-Adapted Combined Rod-Cone B-Wave 0dB Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Combined Rod-Cone B-Wave 0dB Amplitude: Study Eye | -11.5 (24.5) | -44.8 (22.0) | -9.5 (20.0) | 23.0 | -43.0 |
  Dark-Adapted Combined Rod-Cone B-Wave 0dB Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Combined Rod-Cone B-Wave 0dB Amplitude: Fellow Eye | -17.5 (31.4) | -26.0 (21.8) | -6.8 (28.4) | 14.0 | -39.0 |
  Dark-Adapted Combined Rod-Cone A-Wave 11dB Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Combined Rod-Cone A-Wave 11dB Amplitude: Study Eye | 1.3 (34.1) | -29.5 (24.3) | -30.7 (36.3) | -36.5 | -4.5 |
  Dark-Adapted Combined Rod-Cone A-Wave 11dB Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Combined Rod-Cone A-Wave 11dB Amplitude: Fellow Eye | -36.8 (25.0) | -8.5 (8.0) | -3.2 (18.0) | -23.0 | -12.5 |
  Dark-Adapted Combined Rod-Cone B-Wave 11dB Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Combined Rod-Cone B-Wave 11dB Amplitude: Study Eye | -5.0 (34.2) | -26.5 (24.9) | -15.7 (16.5) | -8.0 | -35.0 |
  Dark-Adapted Combined Rod-Cone B-Wave 11dB Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Combined Rod-Cone B-Wave 11dB Amplitude: Fellow Eye | -17.5 (27.4) | -18.8 (20.9) | -15.3 (11.1) | 10.0 | -8.0 |
  Dark-Adapted Oscillatory Potentials Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Oscillatory Potentials Amplitude: Study Eye | -3.5 (2.2) | -12.2 (11.6) | -4.7 (9.4) | -5.0 | -8.0 |
  Dark-Adapted Oscillatory Potentials Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Dark-Adapted Oscillatory Potentials Amplitude: Fellow Eye | -0.3 (3.8) | -6.8 (4.8) | -3.8 (9.5) | -9.0 | -10.5 |
  Light-Adapted Cone B-Wave 0dB Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Light-Adapted Cone B-Wave 0dB Amplitude: Study Eye | -4.7 (6.3) | -4.8 (8.0) | -2.0 (13.9) | 12.5 | -0.5 |
  Light-Adapted Cone B-Wave 0dB Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Light-Adapted Cone B-Wave 0dB Amplitude: Fellow Eye | -4.8 (6.7) | -4.2 (2.4) | 3.3 (25.9) | -5.5 | 9.0 |
  Light-Adapted Cone A-Wave 11dB Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Light-Adapted Cone A-Wave 11dB Amplitude: Study Eye | 1.8 (12.7) | 1.5 (18.2) | -5.5 (13.0) | -10.5 | -2.5 |
  Light-Adapted Cone A-Wave 11dB Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Light-Adapted Cone A-Wave 11dB Amplitude: Fellow Eye | -6.8 (2.4) | -6.2 (3.8) | -1.0 (14.1) | -7.0 | 7.0 |
  Light-Adapted Flicker Amplitude: Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Light-Adapted Flicker Amplitude: Study Eye | -4.5 (11.5) | -10.2 (16.8) | 1.2 (12.8) | -24.0 | -20.0 |
  Light-Adapted Flicker Amplitude: Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Light-Adapted Flicker Amplitude: Fellow Eye | -0.2 (5.3) | -1.8 (11.5) | 3.3 (22.4) | -22.0 | 2.5 |

3. Secondary Outcome: Mean Change in Best Corrected Visual Acuity
Description: Mean change in best corrected visual acuity (BCVA) at Year 2 compared to average of baseline 1 and 2. BCVA is measured via Electronic Visual Acuity (EVA).
Time Frame: Baseline 1 through Year 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters read
Units Other Than Participants: Eyes
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 1 | 0
Number analyzed (Eyes) | 6 | 6 | 6 | 2 | 2 | 0
letters read
  Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Study Eye | 2.7 (3.6) | -0.2 (1.2) | -2.7 (2.5) | -1.0 | -23.0 |
  Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Fellow Eye | -0.2 (2.8) | 0.5 (3.8) | -0.2 (7.6) | -1.5 | -26.0 |

4. Secondary Outcome: Median and Distribution of Change in Best-Corrected Visual Acuity
Description: Median and distribution of change in best-corrected visual acuity (BCVA) at Year 2 compared to average of baseline 1 and 2. BCVA is measured via Electronic Visual Acuity (EVA).
Time Frame: Baseline 1 through Year 2
Population: as for outcome 2
Measure: Median (Full Range); unit: letters read
Units Other Than Participants: Eyes
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 1 | 1 | 0
Number analyzed (Eyes) | 6 | 6 | 6 | 2 | 2 | 0
letters read
  Study Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Study Eye | 4.5 [-2 to 5] | 0.5 [-2 to 1] | -3.0 [-5 to 0] | -1.0 | -23.0 |
  Fellow Eye: number analyzed (Eyes) | 3 | 3 | 3 | 1 | 1 | 0
  Fellow Eye | -1.0 [-3 to 3] | 1.0 [-4 to 4] | -1.5 [-7 to 8] | -1.5 | -26.0 |

5. Secondary Outcome: Formation of Circulating Systemic Anti-AAV or Anti-RS1 Antibodies
Description: Formation of circulating systemic anti-AAV or anti-RS1 antibodies assessed via serologic testing
Time Frame: Day 0 through end of study participation (Year 5 or Year 7)
Population: Includes all participants enrolled in the study and were administered the AAV vector injection, regardless of follow-up.
Measure: Number; unit: events
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 1 | 0
events | 0 | 0 | 0 | 0 | 0 |

6. Secondary Outcome: Change in Retinal Structure as Measured by Optical Coherence Tomography
Description: Change in retinal structure as measured by optical coherence tomography (OCT) compared to average of baseline 1 and 2. Includes a) quantitative measures of total retinal thickness obtained with the Cirrus OCT using macular cube scans, b) qualitative morphologic changes to macula anatomy investigated using the tracking ability of the Heidelberg Spectralis OCT system and c) length of intact ellipsoid zone on the OCT and any findings of restoration of this reflectivity line.
Time Frame: Baseline 1 through end of study participation (Year 5 or Year 7)
Population: Outcome was a secondary outcome. Images were not graded by a Reading Center and therefore data were not collected. Therefore these analyses were not performed.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Change in Central Visual Field Sensitivity as Measured by Microperimetry (MP-1) Visual Field Testing
Description: Change in central visual field sensitivity as measured by microperimetry (MP-1) Visual Field testing compared to average of baseline 1 and 2. Includes mean sensitivities, number of scotomatous points and number of points with a significant change in sensitivity.
Time Frame: Baseline 1 through end of study participation (Year 5 or Year 7)
Population: as for outcome 6
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 0 to end of study participation (Year 5 or Year 7)
Description: All enrolled participants are at risk.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/2 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 2/3 | 0/2 | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 2/2 | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=2) | Cohort 5 (N=1) | Cohort 6 (N=0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=2) | Cohort 5 (N=1) | Cohort 6 (N=0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anterior chamber inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
Central serous chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Halo vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Keratic precipitates (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lacrimal gland enlargement (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Meibomianitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vasculitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subretinal fluid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uveitic glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitritis (Eye disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chorioretinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pilonidal disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Lipids increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Natural progression of disease
Vitreous detachment (Eye disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Natural progression of disease
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Natural progression of disease
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Natural progression of disease
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Natural progression of disease
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Natural progression of disease
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Natural progression of disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT02317887/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT02317887/SAP_001.pdf
  • Informed Consent Form (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT02317887/ICF_002.pdf